CLINICAL TRIAL: NCT04763213
Title: New Predictors in Determining the Need for Invasive Treatment in Non-STEMI During the COVID-19 Pandemic: A Retrospective Study
Brief Title: New Predictors in Determining the Need for Invasive Treatment in Non-STEMI
Acronym: non-STEMI
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ekrem Aksu, Clinical Assis. Prof., MD (Cardiology), Kahramanmaras Sutcu Imam University
Other Study IDs: 05.08.2020-2020/15/10
Record Dates: First submitted 2021-01-29; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Myocard Infarctus
Keywords: Non-ST elevation myocardial infarction acute coronary syndrome; Neutrophil-lymphocyte ratio; Systemic immune inflammation index; Invasive treatment strategy; Conservative strategy
MeSH Terms: interventions — Coronary Angiography; Medical Futility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Invasive treatment: Patients diagnosed with oclusive or nonoclusive coronary artery disease who were treated invasive techniques (Percutaneous Coronary Intervention and Coronary Artery Bypass Grafting)
  Interventions: Diagnostic Test: Coronary Angiography
- Medically treatment: Patients diagnosed with oclusive or nonoclusive coronary artery disease who were treated medically
  Interventions: Diagnostic Test: Coronary Angiography

INTERVENTIONS:
Diagnostic Test: Coronary Angiography — Patients diagnosed with occlusive or nonocclusive coronary artery disease who were treated invasive techniques (Percutaneous Coronary Intervention and Coronary Artery Bypass Grafting)
  Other Names: Invasive treatment
Diagnostic Test: Coronary Angiography — Patients diagnosed with oclusive or nonoclusive coronary artery disease who were treated medically
  Other Names: Medical treatment

SUMMARY:
Non-ST elevation acute coronary syndrome (NSTE-ACS) is a heterogeneous disease with a wide range of treatment options from the medical follow-up to early invasive treatment due to complete occlusion of the culprit artery. Non-ST elevation myocardial infarction acute coronary syndrome (NSTEMI-ACS) is one of the subcomponents of NSTE-ACS, which has an increased mortality rate, and for which early intervention can be vital. Yet, most of these patients require invasive treatment. In fact, some of them are patients who require very early invasive treatment and have a complete occlusion in the culprit artery. Unfortunately, risk scoring systems are not sufficient enough to differentiate these patients. Therefore, the discovery of markers that can be used in the differentiation of NSTEMI-ACS patients with an increased need for invasive treatment and/or complete occlusion of the culprit's vessels, especially during pandemic periods such as the COVID-19 pandemic, has gained importance.

Inflammation is known to play an important role in the etiopathogenesis of coronary artery disease. To the best of our knowledge, there is a lack of literature on the relationship between the need for invasive treatment strategy and/or complete occlusion of the culprit's vessel, and the hematological markers in patients diagnosed with NSTEMI-ACS.

DETAILED DESCRIPTION:
Non-ST elevation acute coronary syndrome (NSTE-ACS) is a heterogeneous disease with a wide range of treatment options from the medical follow-up to early invasive treatment due to complete occlusion of the culprit artery. Non-ST elevation myocardial infarction acute coronary syndrome (NSTEMI-ACS) is one of the subcomponents of NSTE-ACS, which has an increased mortality rate, and for which early intervention can be vital. In the European Society of Cardiology (ESC) guidelines, NSTEMI-ACS is defined as a high-risk condition that requires diagnostic angiography within 2 hours at the latest in those with very high-risk criteria and within 24 hours at the latest in those who do not have high risk. However, the non-invasive approach has come to the fore for the NSTEMI-ACS disease due to the COVID-19 pandemic conditions. In the recently published national consensus report, during the COVID-19 pandemic period, medium-high risk NSTEMI-ACS patients are recommended optimal medical therapy as an alternative treatment method, even if the diagnosis of COVID-19 was excluded, especially in areas where pandemic effects are being experienced intensely. Yet, most of these patients require invasive treatment. In fact, some of them are patients who require very early invasive treatment and have a complete occlusion in the culprit artery. Unfortunately, risk scoring systems are not sufficient enough to differentiate these patients. Therefore, the discovery of markers that can be used in the differentiation of NSTEMI-ACS patients with an increased need for invasive treatment and/or complete occlusion of the culprit's vessels, especially during pandemic periods such as the COVID-19 pandemic, has gained importance.

Inflammation is known to play an important role in the etiopathogenesis of coronary artery disease. In recent years, it has been shown that hematological parameters closely associated with inflammation in people with coronary artery disease may be useful in distinguishing those with increased severity of atherosclerotic involvement and those with high mortality risk. The main markers used in studies are Leukocyte count, neutrophil-lymphocyte ratio (NLR), platelet-lymphocyte Ratio (PLR), systemic immune inflammation index (SII), red blood cell distribution width (RDW), and mean platelet volume (MPV). To the best of our knowledge, there is a lack of literature on the relationship between the need for invasive treatment strategy and/or complete occlusion of the culprit's vessel, and the hematological markers in patients diagnosed with NSTEMI-ACS.

ELIGIBILITY:
Inclusion Criteria:

* NonST elevated myocard ınfarctus
* Elder than 18 years
* Patients who were not have the exclusion criterias

Exclusion Criteria:

* Under the age of 18,
* Recurrent or ongoing chest pain resistant to drug therapy,
* Hemodynamic instability,
* Life-threatening ventricular arrhythmias or cardiac arrest,
* Development of mechanical complications and the presence of dynamic ST-T wave changes (intermittent ST-segment elevation),
* Heart failure,
* Ejection fraction <40,
* Severe anemia,
* Sepsis,
* Malignancy,
* Chronic hematological disease,
* Collagen tissue disease
* Obesity,
* Moderate to severe hepatic failure,
* Renal failure (Glomerular filtration rate <60 ml/min/1.73 m2),
* Severe valvular heart disease,
* Electrolyte disturbance,
* Chronic anti-inflammatory drug use,
* History of chronic inflammatory disease,
* A history of serious infection in the last month
* Patients with missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2018 and December 2019, patients admitted to the Cardiology clinic of a tertiary care hospital with a diagnosis of NSTEMI-ACS were evaluated consecutively
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Predictive factors for Non ST elevated MI Blood prarameters Predictive factors for Non ST eleveted MI | Pretreatment period
  The relationship between inflammation markers such as red cell distribution width (%), mean platelet volume (fL), Systemic immune-inflammation index (platelet count (10^9/L)x neutrophil count (10^9/L)/ lymphocyte count (10^9/L)), neutrophil to lymphocyte ratio (neutrophil count (10^9/L)/ lymphocyte count (10^9/L)), platelet to lymphocyte ratio (neutrophil count (10^9/L)/ lymphocyte count (10^9/L)), and treatment strategy in patients diagnosed with Non-ST myocardial infarction was investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ekrem Aksu, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Collet JP, Thiele H. The 'Ten Commandments' for the 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2020 Oct 1;41(37):3495-3497. doi: 10.1093/eurheartj/ehaa624. No abstract available. PMID 33085966
- [Result] Aktoz M, Altay H, Aslanger E, Atalar E, Aytekin V, Baykan AO, Barcin C, Baris N, Boyaci AA, Cavusoglu Y, Celik A, Cinier G, Degertekin M, Ergonul O, Erturk M, Erol MK, Gorenek B, Gursoy MO, Hunuk B, Kahveci G, Karabay CY, Karaca I, Kayikcioglu M, Keskin M, Kilic T, Kirma C, Kocabas U, Kucukoglu S, Mutlu B, Nalbantgil S, Okuyan E, Okyay K, Kaptan Ozen D, Ozgul S, Ozpelit E, Pirat B, Sert S, Sinan UY, Sener YZ, Tatli E, Tekkesin AI, Tutar E, Ural D, Yildirimturk O. [Consensus Report from Turkish Society of Cardiology: COVID-19 and Cardiovascular Diseases. What cardiologists should know. (25th March 2020)]. Turk Kardiyol Dern Ars. 2020 Mar;48(Suppl 1):1-48. doi: 10.5543/tkda.2020.97198. Turkish. PMID 32250347
- [Result] Sabatine MS, Morrow DA, Cannon CP, Murphy SA, Demopoulos LA, DiBattiste PM, McCabe CH, Braunwald E, Gibson CM. Relationship between baseline white blood cell count and degree of coronary artery disease and mortality in patients with acute coronary syndromes: a TACTICS-TIMI 18 (Treat Angina with Aggrastat and determine Cost of Therapy with an Invasive or Conservative Strategy- Thrombolysis in Myocardial Infarction 18 trial)substudy. J Am Coll Cardiol. 2002 Nov 20;40(10):1761-8. doi: 10.1016/s0735-1097(02)02484-1. PMID 12446059
- [Result] Azab B, Zaher M, Weiserbs KF, Torbey E, Lacossiere K, Gaddam S, Gobunsuy R, Jadonath S, Baldari D, McCord D, Lafferty J. Usefulness of neutrophil to lymphocyte ratio in predicting short- and long-term mortality after non-ST-elevation myocardial infarction. Am J Cardiol. 2010 Aug 15;106(4):470-6. doi: 10.1016/j.amjcard.2010.03.062. PMID 20691303
- [Result] Arbel Y, Finkelstein A, Halkin A, Birati EY, Revivo M, Zuzut M, Shevach A, Berliner S, Herz I, Keren G, Banai S. Neutrophil/lymphocyte ratio is related to the severity of coronary artery disease and clinical outcome in patients undergoing angiography. Atherosclerosis. 2012 Dec;225(2):456-60. doi: 10.1016/j.atherosclerosis.2012.09.009. Epub 2012 Sep 21. PMID 23040448
- [Result] Temiz A, Gazi E, Gungor O, Barutcu A, Altun B, Bekler A, Binnetoglu E, Sen H, Gunes F, Gazi S. Platelet/lymphocyte ratio and risk of in-hospital mortality in patients with ST-elevated myocardial infarction. Med Sci Monit. 2014 Apr 22;20:660-5. doi: 10.12659/MSM.890152. PMID 24751474
- [Result] Sansanayudh N, Anothaisintawee T, Muntham D, McEvoy M, Attia J, Thakkinstian A. Mean platelet volume and coronary artery disease: a systematic review and meta-analysis. Int J Cardiol. 2014 Aug 20;175(3):433-40. doi: 10.1016/j.ijcard.2014.06.028. Epub 2014 Jun 28. PMID 25017904
- [Result] Isik T, Uyarel H, Tanboga IH, Kurt M, Ekinci M, Kaya A, Ayhan E, Ergelen M, Bayram E, Gibson CM. Relation of red cell distribution width with the presence, severity, and complexity of coronary artery disease. Coron Artery Dis. 2012 Jan;23(1):51-6. doi: 10.1097/MCA.0b013e32834e4f5c. PMID 22133925
- [Result] Yang YL, Wu CH, Hsu PF, Chen SC, Huang SS, Chan WL, Lin SJ, Chou CY, Chen JW, Pan JP, Charng MJ, Chen YH, Wu TC, Lu TM, Huang PH, Cheng HM, Huang CC, Sung SH, Lin YJ, Leu HB. Systemic immune-inflammation index (SII) predicted clinical outcome in patients with coronary artery disease. Eur J Clin Invest. 2020 May;50(5):e13230. doi: 10.1111/eci.13230. Epub 2020 May 11. PMID 32291748